CLINICAL TRIAL: NCT04317196
Title: Molecular Epidemiology Study of the Association of Copy Number Variations in the SMN Genes With Acute Kidney Injury After Heart Surgery
Brief Title: Association of Copy Number Variations in the SMN Genes With Acute Kidney Injury After Heart Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XHEC-C-2019-111
Record Dates: First submitted 2019-11-26; First posted 2020-03-23 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-07

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective cohort study aims to explore the susceptibility to acute kidney injury after heart surgery in SMN1+/- genotype population. This study also aims to analysis the effect of SMN1+/- genotype on postoperative AKI and the development of chronic kidney disease, as well as dose-compensating effect of different copy number of SMN2 gene on SMN1 +/- genotype.

DETAILED DESCRIPTION:
This prospective cohort study aims to explore the susceptibility to acute kidney injury after heart surgery in SMN1+/- genotype population. Real-time PCR is used to detect copy number variations in the peripheral blood SMN gene on 1206 patients with heart surgery. This study also aims to analysis the effect of SMN1+/- genotype on postoperative AKI and the development of chronic kidney disease, as well as dose-compensating effect of different copy number of SMN2 gene on SMN1 +/- genotype.

ELIGIBILITY:
Inclusion Criteria:

* Age: Children (1 month -17 years old) and adults (18-80 years old);
* Sex: All;
* Those who will receive selective cardiac surgery with cardiopulmonary bypass;
* Those who signed the informed consent.

Exclusion Criteria:

* Those with glomerular filtration rate: eGFR<15ml/min/1.73m2, and those who have received the renal replacement therapy before surgery;
* Those who have received nephrectomy and kidney transplantation;
* Those who have suffered from AKI before;
* Those with incomplete medical history or clinical data.

Ages: 1 Month to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Sampling Method: Non-Probability Sample
Enrollment: 1206 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with occurrence of acute kidney injury (AKI) after cardiac surgery | 48 hours
  The definition of the occurrence of acute kidney injury is according to the acute kidney injury (AKI) definition and staging criteria released by Kidney Disease: Improving Global Outcomes (KDIGO) in the year 2012

SECONDARY OUTCOMES:
Number of participants with occurrence of acute kidney disease (AKD) after cardiac surgery | 3 months
  The definition of the occurrence of acute kidney disease is according to the acute kidney disease (AKD) definition criteria released by Kidney Disease: Improving Global Outcomes (KDIGO) in the year 2012
Glomerular Filtration Rate(GFR) | 90 days
  Glomerular filtration rate (GFR) is defined as the volume of plasma that is filtered by the glomeruli per unit of time, and is usually measured by estimating the rate of clearance of a substance from the plasma.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China